CLINICAL TRIAL: NCT00285298
Title: Pentoxifylline and Progression of Chronic Kidney Disease in Moderate-to-high Risk Patients: a Pilot Randomized, Placebo-controlled, Double-blind Trial.
Brief Title: Pentoxifylline and Progression of Chronic Kidney Disease in Moderate-to-high Risk Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Robert M. Perkins, MD, Geisinger Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-11010(1); 11010A (NKF)
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2009-09

CONDITIONS: Kidney Failure, Chronic
Keywords: proteinuria; Kidney failure, chronic
MeSH Terms: conditions — Kidney Failure, Chronic; Proteinuria | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pentoxifylline (Experimental)
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline
  Arms: Pentoxifylline
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the investigators study is to assess the impact of therapy with Pentoxifylline (PTF), a nonspecific phosphodiesterase inhibitor, on kidney function in patients at high-risk for progression to end-stage renal disease. The investigators hypothesize that therapy with Pentoxifylline will slow progression of kidney disease over time.

DETAILED DESCRIPTION:
The treatment objective for chronic kidney disease (CKD), regardless of etiology, is to slow or halt progression of renal dysfunction and reduce proteinuria (in those patients with proteinuric renal disease). Multi-drug medical regimens remain the cornerstone of therapy for medical-renal disease, often with an angiotensin converting enzyme inhibitor and/or an angiotensin receptor blocker. These therapies, though often efficacious, have not been shown to halt disease progression entirely, and the medical therapy of renal disease remains suboptimal.

PTF is a safe, generally well-tolerated drug currently indicated for symptomatic and functional relief of intermittent claudication presumed due to chronic occlusive arterial disease of the limbs. A number of small studies in patients across a range of renal disease states show that PTF can reduce proteinuria, an important component of treatment of CKD. It is not known, however, if the drug will slow progression of CKD as measured by glomerular filtration rate.

Comparisons: subjects randomized to receive PTF compared with those randomized to receive placebo

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years of age or older currently being treated with an ACE-I or ARB and with one of the following conditions:

1. Non-nephrotic range proteinuria (between 1 and 3 grams/day by 24-hr collection), hypertension (blood pressure >130/80 or current use of antihypertensive drug therapy), and an eGFR of less than or equal to 40 ml/minute but greater than 20 ml/minute.

   OR
2. Nephrotic range proteinuria (>=3 grams/day proteinuria) by 24-hr urine collection, and an eGFR greater than 20 ml/minute

Exclusion Criteria:

1. Acute renal failure: defined by >25% decrease in eGFR over one month
2. Pregnancy or currently breast-feeding
3. Current use of cytotoxic drug therapy (cyclophosphamide, cyclosporine, mycophenolate mofetil, prednisone, chlorambucil) or a current indication for, and plan to implement, such therapy.
4. Current use of PTF
5. Contraindication to use of PTF drug: history of PTF or theophylline allergy, history of severe retinal hemorrhage or recent cerebral hemorrhage
6. Current use of theophylline
7. Contraindication to ACE-I or ARB.
8. Fewer than 2 measured serum creatinine values separated by 6 months prior to potential enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Rate of decline in estimated glomerular filtration rate over one year | 1 year

SECONDARY OUTCOMES:
50% reduction in proteinuria | 1 year
Change in slope of 1/serum creatinine vs time | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Perkins, MD, Study Director — Walter Reed Army Medical Center, Nephrology Service

REFERENCES:
- [Result] Perkins RM, Aboudara MC, Uy AL, Olson SW, Cushner HM, Yuan CM. Effect of pentoxifylline on GFR decline in CKD: a pilot, double-blind, randomized, placebo-controlled trial. Am J Kidney Dis. 2009 Apr;53(4):606-16. doi: 10.1053/j.ajkd.2008.11.026. Epub 2009 Feb 12. PMID 19216016
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745